CLINICAL TRIAL: NCT01847898
Title: Study to Evaluate the Clinical Performance of the VBS System for the Treatment of Osteoporotic Vertebral Fractures in a Multicenter, Randomized, Controlled Setting
Brief Title: Study on the Treatment of Osteoporotic Vertebral Fractures Using Vertebral Body Stenting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Synthes GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU-SPI-S-06-134-01; STU-SPI-S-06-134-01 (Other: Synthes GmbH)
Record Dates: First submitted 2009-08-27; First posted 2013-05-07 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Vertebral Body Fractures
Keywords: Osteoporosis; Vertebral Body; Compression Fracture; Kyphoplasty
MeSH Terms: conditions — Osteoporosis; Fractures, Compression | interventions — Kyphoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vertebral Body Stenting (VBS) (Experimental)
  Interventions: Procedure: Vertebral Body Stenting (VBS)
- Balloon Kyphoplasty (Experimental)
  Interventions: Procedure: Balloon Kyphoplasty

INTERVENTIONS:
Procedure: Vertebral Body Stenting (VBS) — Vertebral Augmentation with a Stent
  Arms: Vertebral Body Stenting (VBS)
Procedure: Balloon Kyphoplasty — Vertebral Augmentation with a Balloon (device not specified)
  Arms: Balloon Kyphoplasty

SUMMARY:
This is a randomized, controlled study to document and evaluate the clinical performance of the Vertebral Body Stenting (VBS) System in osteoporotic fractures of the thoracic and lumbar spine.

The randomized, controlled trial (RCT) will compare patients with VBS and Balloon Kyphoplasty.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 50
2. 1 to 3 contiguous target vertebral compression fractures (VCF) meeting the following criteria:
3. Fracture due to diagnosed or presumed underlying primary or secondary osteoporosis (Patients with AO type A1.x fractures and A3.1 fractures may be included in the study).
4. All target VCFs are between Th5 and L5

   * All target VCFs to be treated show either:

     * Height change: An acute (< 6 month) change in VB height (>15% height loss) with height loss at the anterior, middle or posterior portion of the VB consistent with a worsening of 1 or more grades by the Genant criteria, OR
     * Positive MRI or bone scan: VB shows hyperintense signal on MRI-T2 or STIR sequence or target VB is positive on radionuclide bone scan
   * Back pain correlating with the location of at least one VCF
5. Treatment of all target VCFs is technically feasible by and clinically appropriate for BOTH vertebroplasty and balloon kyphoplasty
6. No major surgery to the spine planned for at least 1 month following enrollment
7. Pre-treatment back pain by numerical rating scale (NRS) score >= 4 (0-10 scale)
8. Subject is able to understand the risks and benefits of participating in the study and is willing to provide written informed consent
9. Psychosocially, mentally and physically able to fully comply with the protocol requirements for the duration of the study including adhering to scheduled visits, treatment plan, completing forms and other study procedures

Exclusion Criteria:

1. VB morphology or configuration is such that either balloon kyphoplasty OR vertebroplasty is not technically feasible for the targeted VCFs
2. Fracture due to high-energy trauma
3. Suspected OR proven cancer inside index vertebral body.
4. Disabling back pain due to causes other than acute fracture (e.g., sacroiliac fracture, symptomatic degenerative disc disease, lumbar spinal stenosis)
5. Any painful VCF with fracture age > 6 months
6. Patients with primary tumors of the bone (e.g., osteosarcoma) or solitary plasmacytoma at site of the index VCF. Patients with these tumors in anatomic sites other than the index VCF are eligible.
7. Any objective evidence of neurologic compromise at baseline
8. Previous balloon kyphoplasty or vertebroplasty for any VCF
9. Spine stabilization beyond balloon kyphoplasty or vertebroplasty required for targeted VCFs
10. Significant clinical comorbidity that may potentially interfere with long-term data collection or follow-up (e.g., dementia, severe comorbid illness)
11. Patients requiring the use of high-dose steroid (>= 100mg prednisone or 20 mg dexamethasone per day), IV pain medication, or nerve block to control chronic back pain unrelated to index VCF(s). Patients who receive high-dose steroids for treatment of their cancer (for at least 30 days) are eligible.
12. Patients who may require allogeneic bone marrow transplantation during the course of the study
13. Spinal cord compression or canal compromise requiring decompression
14. Patients with osteoblastic tumors at the site of index VCF. Patients with osteoblastic tumors of vertebral levels not intended for kyphoplasty may be enrolled.
15. MRI contraindication (e.g. cerebral aneurysm clips, pacemaker, implanted biostimulators, cochlear implants, penile prosthesis)
16. Spinal instability as indicated by neurologic deficit, kyphosis >30°, compression >50%, translation > 4 mm, interspinous-process widening.
17. Pre-existing conditions contrary to either balloon kyphoplasty or vertebroplasty, such as:

    * Irreversible coagulopathy or bleeding disorder. Note regarding reversible coagulopathies: Subjects on coumadin or other anticoagulants may participate. Investigators should follow routine practices for perioperative discontinuation and re-initiation of anticoagulants.
    * Allergy to any device materials (e.g., bone cement) for balloon kyphoplasty or vertebroplasty. Note that in subjects with allergy to iodine-based contrast, other non-iodine contrast solutions may be used.
    * Any evidence of VB or systemic infection
18. Pregnant or child-bearing potential

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-09-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Increase and maintenance of the vertebral body height | 12 months
  The anterior edge, mid height and posterior edge of the index vertebral body are measured pre-operatively standing, after prone intraoperative positioning on the table (dynamic fracture mobility), intra-operatively following balloon dilation (height restoration), after balloon deflation and removal, after cement deposition, and finally postoperative standing. Anterior, middle and posterior height measurements will be made at each time-point during the study to measure maintenance of vertebral body height over time. The ratio between anterior and mid or posterior edge height (Beck-index) is calculated to avoid the problem of image calibration. In addition, the relative height fractions in comparison to the nearest healthy vertebral body (referent level) are calculated. Finally, local and regional sagittal angles and overall lumbar lordosis or thoracic kyphosis, respectively, are assessed for measurement of improvement of alignment.
Visual analog scale (VAS) for back pain | 12 months
  Pain assessment by the patients using the VAS back pain from 0 to 10. In this scale 0 means "no pain" and 10 is the "worst pain imaginable". A pre- to postoperative difference of at least 2 observed during the course of the therapy is regarded as clinically relevant.
Adverse events | 12 months
  * Any re-operations, revisions, and removals or supplemental fixation at the index level(s) is considered a study failure.
  * Any intra-operative system malfunction, misplacement of the balloon or stent, balloon or stent fracture, or failure of the balloon or stent to fully deploy is considered a study failure.

SECONDARY OUTCOMES:
Radiographic evaluations | 2 years
  Evaluation of osteolysis surrounding the VBS System and/or cement; Evaluation of adjacent level arthritis; Evaluation of bridging trabecular bone at intradiscal spaces adjacent to the treated level(s); Assessment of segmental kyphosis/lordosis at the treated and adjacent level(s) Evaluation of all vertebral body fractures directly above and below the treated level(s
Global assessment by the patient using the VAS | 2 years
  Patients globally assess their overall satisfaction with the treatment using the VAS, where 0 = totally dissatisfied and 10 = totally satisfied. A six-level question comparing the current situation to the preoperative state of health is also used.
VAS leg pain | 2 years
  VAS leg pain from 0 to 10. In this scale 0 means "no pain" and 10 is the "worst pain imaginable".
Analgesic usage | 2 years
  Analgesic consumption is documented in the categories - none, Paracetamol (Acetaminophen), Nonsteroidal anti-inflammatory drugs (NSAID), Metamizole, mild opiates and strong opiates at baseline and each follow-up office visit. This information is obtained with the help of medical staff or the patient's family and relatives.
Neurological assessment of root tension signs, muscle strength, sensory deficit and reflexes | 2 years
  Assessment of root tension signs (yes/no), muscle strength (normal/decreased), sensory deficit (yes/no) and reflexes (normal/decreased/increased) will be conducted at baseline and each follow-up visit
Symptoms associated with position/direction of cement extrusion | 2 years
  Symptoms associated with position/direction of cement extrusion: epidural, pulmonary, intradiscal, large vessels, foraminal, paraspinal soft tissue, paravertebral vessels, other.
Disability using the Oswestry Disability Index (ODI) | 2 years
  Oswestry Disability Index (ODI), version 2.1 will be used.
Quality of Life Evaluation using the EuroQol, general quality of life questionnaire (EQ-5D) | 2 years
  The EQ-5D (EuroQol, general quality of life questionnaire) will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Paul F. Heini, Prof. Dr. med., Principal Investigator — Klinik Sonnenhof, Bern, Switzerland
Locations (5):
- Austria (2):
  - Universitätsklinik für Unfallchirurgie, Graz
  - AKH, Vienna
- Germany (3):
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Universitätsklinikum, Münster
  - Universitätsklinik und Poliklinik für Chirurgie, Rostock